CLINICAL TRIAL: NCT03344432
Title: Correlation of Intraocular Pressure With Intracranial Pressure in Childs With Severe Trauma Brain Injury
Brief Title: Correlation Intraocular Pressure With Intracranial Pressure
Acronym: IOPICPTBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, KARLA ISIS AVILES MARTINEZ, Dra. Karla Isis Avilés-Martínez, Hospital Civil de Guadalajara
Other Study IDs: HCG/CI-0693/15
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Intraocular Pressure; Intracranial Pressure Increase; Trauma, Brain; Children, Only
MeSH Terms: conditions — Intracranial Hypertension; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- With intraocular pressure high: Intracranial pressure equal or more than 20 mmHg
  Interventions: Diagnostic Test: with intraocular pressure high; Diagnostic Test: without intraocular pressure high
- Without intraocular pressure high: Intracranial pressure smaller than 20 mmHg
  Interventions: Diagnostic Test: with intraocular pressure high; Diagnostic Test: without intraocular pressure high

INTERVENTIONS:
Diagnostic Test: with intraocular pressure high — Measurement of intraocular pressure The measurement will be made with a electronic minimum contact tonometer for measuring intraocular pressure immediately before the placement of the invasive catheter for measurement of intracranial pressure.
Diagnostic Test: without intraocular pressure high — Measurement of intraocular pressure The measurement will be made with a electronic minimum contact tonometer for measuring intraocular pressure immediately before the placement of the invasive catheter for measurement of intracranial pressure.

SUMMARY:
Severe Trauma Brain Injury (TBIs) is a public health problem and monitoring of Intracranial Pressure (ICP) is a determinant key of it prognosis. Within the noninvasive methods to estimate the ICP, the measurement of intraocular pressure has been proposed because of its biological plausibility (proximity of the eye to the encephalic contend).

Objective. Correlate intraocular pressure with ICP in children with TBIs and obtain their utility values.

DETAILED DESCRIPTION:
Severe Trauma Brain Injury (TBIs) is a public health problem and monitoring of Intracranial Pressure (ICP) is a determinant key of it prognosis. Within the noninvasive methods to estimate the ICP, the measurement of intraocular pressure has been proposed because of its biological plausibility (proximity of the eye to the encephalic contend).

Objective. Correlate intraocular pressure with ICP in children with TBIs and obtain their utility values.

Material and methods. Correlation and diagnostic test design study. Inclusion criteria: children with TBIs admitted to the emergency room and indication of catheter for ICP measurement.

Exclusion criteria: injury or ophthalmic disease, glaucoma, encephalic death. Intraocular pressure was measured with electronic tonometer in both eyes prior to placement of the catheter for ICP measurement.

Correlation was estimated with Spearman's Rho. The utility values of the diagnostic test were obtained from an Receiver Operating Characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

1. Children with severe trauma brain injury (Coma Glasgow Scale smaller than 9 points),
2. who have been admitted to the pediatric emergency room
3. and in whom the treating neurosurgeon has decided to place a catheter for intracranial pressure measurement.

Exclusion Criteria:

1. Ocular trauma,
2. brain death,
3. know eye disease,
4. refusal of parents or guardians to participate in the study.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children of 2 at 15 years old with severe trauma brain injury (Coma Glasgow Scale smaller than 9 points), in pediatric emergency room, with indication by the neurosurgeon to place a invasive catheter for intracranial pressure measurement.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure smaller than 20 mmHg | Immediately
  Abscence of increased intraocular pressure (smaller than 20 mmHg) without intracranial pressure smaller than 20 mmHg.

SECONDARY OUTCOMES:
Intraocular pressure equal or more than 20 mmHg | Immediately
  Intraocular pressure equal or more than 20 mmHg with Intracranial pressure equal or more than 20 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Karla Isis I Aviles Martinez, PhD, Principal Investigator — Hospital Civil Fray Antonio Alcalde
Locations (1):
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided